CLINICAL TRIAL: NCT04734834
Title: Clinical Study On "Prodovite®" In Athletic Performance
Brief Title: Efficacy Of "Prodovite®" In Athletic Performance
Acronym: VMP35SPORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Victory Nutrition International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VNI-VMP35SPORTS-OCT2019 2020R1; VMP35 (Registry Identifier: VNI Inc)
Record Dates: First submitted 2020-10-10; First posted 2021-02-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: SPORTS NUTRITION
Keywords: "Prodovite®" VMP35; 90-Day; 150 Subjects; Double-Blind, Placebo-Control Study; Endurance Athletic Performance; Adverse Events Monitoring

STUDY DESIGN:
Intervention Model Description: A double-blind placebo-controlled investigation to evaluate the efficacy of "Prodovite®" VMP35 in Boosting Athletic Performance in Athletes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind placebo-controlled investigation in 150 subjects,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be provided orally to the Placebo Group. Placebo will be blinded and labeled either as "A" or "B".
  Interventions: Dietary Supplement: "Prodovite®" VMP35
- "Prodovite®" VMP35 (Active Comparator): "Prodovite®" VMP35 will be provided orally to the Treatment Group. "Prodovite®" VMP35 will be blinded and labeled either as "A" or "B".
  Interventions: Dietary Supplement: "Prodovite®" VMP35

INTERVENTIONS:
Dietary Supplement: "Prodovite®" VMP35 — Efficacy of "Prodovite®" VMP35 will be Assessed as Compared to Placebo

SUMMARY:
A novel patent-pending "Prodovite®" VMP35 Multi-Nutrient-Complex (MNC), a vitamin, mineral, and phytonutrient encapsulated liquid formulation, was prepared using a novel proprietary SK713 SLP multi-lamellar non-GMO phospholipid nutrient absorption/delivery technology in a state-of-the-art multistep cGMP and NSF-certified manufacturing facility. This developmental technology is biodegradable and biocompatible. Preliminary study in our laboratory demonstrated the efficacy of "Prodovite®" VMP35 in Sports Nutrition. The investigators hypothesize that "Prodovite®" VMP35 supplement will enhance strength, endurance, and athletic performance; and improve energy output, lean-body muscle mass, increase exercise tolerance, recovery, and improve anabolic parameters in healthy human subjects. The aim of this randomized double-blind placebo-controlled study is to evaluate the effect of oral supplementation of "Prodovite®" VMP35 on the parameters. The investigators hypothesize that "Prodovite®" VMP35 supplementation will enhance all the athletic parameters and improve blood chemistry parameters in healthy human subjects. Accordingly, 150 healthy male and female subjects will be randomly assigned to receive either "Prodovite®" VMP35 or placebo in the form of single dose sealed containers for 90 consecutive days and muscle strength, endurance, speed, anabolic/catabolic parameters and muscle mass will be evaluated by dual energy X-ray absorptiometry (DEXA), hand-grip strength test, cycle ergometer test, spirometer assessment and assay of Blood chemistry and serum biomarkers will be evaluated before and after intervention.

DETAILED DESCRIPTION:
Higher level athletic performance induces greater demands on nutrient and oxygen utilization and hydration. Consistent performance-induced chronic resource depletion from demands of this level can induce an increasing anaerobic, hypoxic/acidic environment, promoting anaerobic metabolic events (i.e. anaerobic glycolysis). Disorders arising from this depletion include chronic inflammation, cramps, and pain, and induce a defensive expenditure of alkalinizing buffers in hemoglobin (i.e. histidine), to prevent a dangerous lowering of blood pH. The physical demands of higher levels of athletic performance deplete biological resources predisposing a greater incidence of chronic problems such as cramps, inflammation, muscle injury and pain. A Phase 1 Pilot Validation Study was conducted in three healthy young trained male athletes (Age: 32-39 years) over a period of 90 consecutive days, with a 2-week intermediate evaluation1. Subjects consumed 30 mL (1-ounce) of "Prodovite®" VMP35, a World Anti-Doping Association (WADA) compliant iron-free liquid "Prodovite®" VMP35 vitamin, mineral and phytonutrient complex (MNC) on an empty stomach before engaging in a rigorous exercise regimen in the morning. They consumed another ounce of the "Prodovite®" VMP35 again mid-afternoon of the same day. Total blood chemistry including free and bound testosterone levels, as well as changes in their exercise performance activities were closely monitored and recorded prior to consuming the "Prodovite®" VMP35, during the intermediate 2-week evaluation, and then again at the end of the study period. In the 2-week Phase 1 evaluation, 1 ounce of "Prodovite®" VMP35 taken within 30 minutes before engaging in a rigorous exercise regimen, induced dramatic improvements in athletic exercise performance. Following "Prodovite®" VMP35 supplementation, physiological health including physical strength, stamina, respiratory parameters, energy level, and sleep quality increased, and blood chemistry parameters were improved. Before "Prodovite®" VMP35 intake, one subject was struggling with 270 lbs. for 4 reps on the banded reverse Hack Squat, while after supplementation, subject achieved 270 lb.s for 10 reps; rested, then the very next set increased to 320 lbs. for 10 reps. The set after that (the 3rd and final set of that exercise), weight increased again to 360 lbs. for 8 reps. In another subject on the same equipment, pre-"Prodovite®" VMP35 supplementation, the squat result was 405 lbs. for 10 reps, while post-"Prodovite®" VMP35 supplementation, the squat increased significantly to 455 lbs. for 6 reps. Pre-"Prodovite®" VMP35 intake, one exercise in particular, the subject was able to perform the banded reverse hack squat with 160 lbs for one set of 8 reps. After "Prodovite®" VMP35 intake, the subject increased squat performance to 180 lbs. for 2 sets of 10 reps. On the Hammer Strength banded incline chest press, pre-"Prodovite®" VMP35, subject's working weight sets were 160 lbs. Post-"Prodovite®" VMP35 sets increased to 180 lbs. Another increase in strength was experienced in banded Hammer Strength incline press. Pre-VMP35, Subject was doing 180 lbs. for 10 reps, which was increased to 230 lbs. for 10 reps post "Prodovite®" VMP35. On side lateral dumbbell raises subject's working weight increased from 20 lbs. Pre-"Prodovite®" VMP35 to 25 lbs. Post- Prodovite® VMP35 supplementation, subjects were able to push a little harder and achieve extra reps with shorter rest periods. Overall, a significant increase in strength was noticed in all subjects and all subjects experienced shorter recovery time between sets and post-workout. Based on these encouraging data, investigators propose to conduct the following full-blown investigation. This pilot investigation inspired our team to conduct a randomized placebo-controlled, double-blind investigation in 150 volunteers (age: 18-74 years) over a period of 90 consecutive days. A statistician will be involved in this project. Body weight, body mass index (BMI), waist circumference, blood chemistry, blood pressure and heart rate, body and hand grip strength, speed and endurance studies including open circuit spirometry-based assessment of pulmonary function will be assessed. Other parameters to be evaluated include oxygen consumption, CO2 production and metabolic parameters, VO2 max, respiratory exchange ratio (RER), anaerobic threshold, ventilatory equivalents for oxygen (VE/V02) and exhaled carbon dioxide (VE/VC02). Subjects will participate in completed maximal graded exercise tests (GXT) on a treadmill or in set distance open-field sprints using open-circuit spirometry. Lower and Upper Body Strength will be evaluated. E-Diary will be provided to all participants. Survey Monkey program will be provided to all subjects and regularly updated by all study participants daily and endorsed by the Principal Investigator and Sub-Investigators.

ELIGIBILITY:
Inclusion criteria

1. Agrees to written as well as audio-visual informed consent
2. Ability to understand the risks/benefits of the study protocol
3. Healthy male and female, human subjects 18-74 years of age
4. Subjects experienced with at least six months of regular athletic performance training

Exclusion criteria

1. Uncooperative Subjects
2. Subjects with chronic illness (diabetes, cardiovascular disease, cancer, arthritis, etc) or those on prescription medication excluded (except for birth control pills)
3. Any conditions that prevent the subject from participating in physical activities.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — A Total of 150 Healthy Male and Female Subjects (50:50) will be recruited after rigorous Evaluation
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Body Weight (Kg) | Over the period of 90 consecutive days
  Body Weight (Kg) will be measured in both placebo and "Prodovite®" groups
Height (m) | Over the period of 90 consecutive days
  Height (m) will be measured in both placebo and "Prodovite®" groups
Body Mass Index (kg/m^2) | Over the period of 90 consecutive days
  Body Mass Index (kg/m^2) will be measured in both placebo and "Prodovite®" groups
Body circumference (in cm) | Over the period of 90 consecutive days
  Body Circumference [arm (cm)], [waist (cm)], [hip (cm)], and [calf (cm)] will be measured in both placebo and "Prodovite®" groups
Waist Hip Ratio | Over the period of 90 consecutive days
  Waist Hip Ratio will be measured in both placebo and "Prodovite®" groups
Knee-Heel Length (cm) | Over the period of 90 consecutive days
  Knee-Heel Length (cm) will be measured in both placebo and "Prodovite®" groups
Blood Pressure (mm Hg) | Over the period of 90 consecutive days
  Blood Pressure including Systolic (mm Hg) and Diastolic Blood pressure (mm Hg) will be measured in both placebo and "Prodovite®" groups
Total Cholesterol (mg/dL) | Over the period of 90 consecutive days
  Total Cholesterol (mg/dL) in both placebo and "Prodovite®" groups
Total Testosterone (ng/dL) | Over the period of 90 consecutive days
  Total Testosterone (ng/dL) in both placebo and "Prodovite®" groups
Percent Body Fat (%) | Over the period of 90 consecutive days
  Percent Body Fat (%) Measurement by Dual Energy X-Ray Absorptiometry (DEXA) in both placebo and "Prodovite®" groups
Bone Mineral Density (g/cm2) | Over the period of 90 consecutive days
  Bone Mineral Density (g/cm2) Measurement by Dual Energy X-Ray Absorptiometry (DEXA) in both placebo and "Prodovite®" groups
Fat Free Mass [Body fat percent (%) x scale weight = fat mass] | Over the period of 90 consecutive days
  Fat Free Mass [Body fat percent (%) x scale weight = fat mass] Measurement by Dual Energy X-Ray Absorptiometry (DEXA) in both placebo and "Prodovite®" groups
Lean Body Mass (lbs)[scale weight - fat mass = lean body mass] | Over the period of 90 consecutive days
  Lean Body Mass (lbs)[scale weight - fat mass = lean body mass] Measurement by Dual Energy X-Ray Absorptiometry (DEXA) in both placebo and "Prodovite®" groups
In-Body Electrical Impedance Value | Over the period of 90 consecutive days
  Body Composition Analysis (In-Body Electrical Impedance) in both placebo and "Prodovite®" groups
Hand-Grip Strength (lb) | Over the period of 90 consecutive days
  Digital Hand Dynamometer will be used for assessing Hand-Grip Strength (lb) [Percent (%) Change] in both placebo and "Prodovite®" groups
Strength Assessment (lb/reps) | Over the period of 90 consecutive days
  Maximum Push-Up Test for Assessing Upper Body Strength (lb/reps) in both placebo and "Prodovite®" groups
Maximum Power Output (W) (as part of Endurance Assessment) | Over the period of 90 consecutive days
  A Cycle Ergometer will be used for measuring Maximum Power Output (W) in both placebo and "Prodovite®" groups
VO2 Max (L.Min-1) (as part of Endurance Assessment) | Over the period of 90 consecutive days
  A Cycle Ergometer will be used for measuring VO2 Max (L.Min-1) in both placebo and "Prodovite®" groups
Respiratory Exchange Ratio (RER) (as part of Endurance Assessment) | Over the period of 90 consecutive days
  A Cycle Ergometer will be used for measuring Respiratory Exchange Ratio (RER) in both placebo and "Prodovite®" groups

SECONDARY OUTCOMES:
Study Compliance | Over the period of 90 consecutive days
  Study Compliance including subject drop-outs and recording of supplement intake will be critically evaluated in Both Placebo- and "Prodovite®" Groups
Adverse Events Monitoring | Over the period of 90 consecutive days
  Adverse Events including headache, nausea, vomiting, diarrhea, rash, fever, muscle cramp and weight gain will be critically Monitored in Both Placebo- and "Prodovite®" Groups

CONTACTS AND LOCATIONS:
Overall Officials: BRUCE S MORRISON, DO, Principal Investigator — Medical Director, SPORTS MEDICINE & FAMILY PHYSICIAN, HUNTINGDON VALLEY, PA 19006; Jeffrey M Galvin, MD, Study Director — Medical Director, Vitality Medical Wellness Institute, Charlotte, NC; Terrance Shane (Bear) Robinson, MS, Study Director — Director, Hardcore Serious Fitness. Huntersville, NC
Locations (2):
- United States (2):
  - Vitality Medical Wellness Institute, 9350 Benfield Road, Suite #110, Charlotte, North Carolina
  - Hardcore Serious Fitness, 13730 Statesville Road, Huntersville, North Carolina

IPD SHARING:
Plan to Share IPD: No
This is a double-blind placebo-controlled study. Confidentiality will be strictly Maintained. No Participant's name will be disclosed. All Data will be Kept with the Principal Investigator Under Lock & Key

REFERENCES:
- [Result] Corbier JR, Downs BW, Kushner S, Aloisio T, Bagchi D, Bagchi M. VMP35 MNC, a novel iron-free supplement, enhances cytoprotection against anemia in human subjects: a novel hypothesis. Food Nutr Res. 2019 May 9;63. doi: 10.29219/fnr.v63.3410. eCollection 2019. PMID 31105509